CLINICAL TRIAL: NCT03874195
Title: Usability Testing of a Web-based Tool to Prepare Patients for Palliative Care
Brief Title: Palliative Care For Me (PCforMe)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00075906
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Palliative Care

STUDY DESIGN:
Intervention Model Description: The Investigator will 1:1 randomize patients to an Active Control arm or Intervention arm. Both arms will receive a tablet computer (iPad or Galaxy Tab based on preference) connected to the internet with disposable headphones to use for up to 30 minutes. Subjects in the Active Control arm will receive a list of three nationally-recognized websites to receive information on palliative care - www.palliativedoctors.org; getpalliativecare.org; and Wikipedia "Palliative Care" https://en.wikipedia.org/wiki/Palliative_care). Intervention Arm subjects will receive access to PCforMe.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Subjects in the Active Control arm will receive a list of three nationally-recognized websites to receive information on palliative care - www.palliativedoctors.org; getpalliativecare.org; and Wikipedia "Palliative Care" https://en.wikipedia.org/wiki/Palliative care).
  Interventions: Behavioral: Access to three nationally-recognized Palliative Care websites for review
- Intervention (Experimental): Intervention Arm subjects will receive access to PCforMe.
  Interventions: Behavioral: Access to PCforMe for review

INTERVENTIONS:
Behavioral: Access to PCforMe for review — Intervention Arm subjects will receive access to PCforMe.
  Other Names: Knowledge of Palliative Care; Prepartion for Palliative Care appointment; Confidence in Palliative Care discussion with provider
  Arms: Intervention
Behavioral: Access to three nationally-recognized Palliative Care websites for review — Subjects in the Active Control arm will receive a list of three nationally-recognized websites to receive information on palliative care
  Other Names: Knowledge of Palliative Care; Prepartion for Palliative Care appointment; Confidence in Palliative Care discussion with provider
  Arms: Control

SUMMARY:
The purpose of this study is to test the usability of PCforMe, a web-based preparation and engagement tool about palliative care, during a pre-visit pilot trial in outpatient palliative care at the Duke Cancer Institute Palliative Care Clinic.

DETAILED DESCRIPTION:
The Investigator will 1:1 randomize patients to an Active Control arm or Intervention arm. Both arms will receive a tablet computer (iPad or Galaxy Tab based on preference) connected to the internet with disposable headphones to use for up to 30 minutes. Subjects in the Active Control arm will receive a list of three nationally-recognized websites to receive information on palliative care - www.palliativedoctors.org; getpalliativecare.org; and Wikipedia "Palliative Care" https://en.wikipedia.org/wiki/Palliative_care). Intervention Arm subjects will receive access to PCforMe.

PCforMe is an online, web-based, interactive tool to prepare patients for a clinical palliative care encounter. PCforMe is accessible through www.pcforme.org. It does not collect any patient information, including identifiers (e.g. name, email address, disease, location) or health information (e.g. disease, symptom severity or location). The system uses a combination of animated videos and user-answered questions to generate a "Palliative Care Passport", which is a summary of information entered into the system. Research staff will print out the Passport for patients and hand it to them prior to the appointment.

Queries for users include standard-of-care questions asked by palliative care clinicians, including areas that patients want to more learn about. No diagnoses, medication advice, or clinical assessments are made or given.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants will be identified by reviewing clinic appointment listings in EPIC (e.g., diagnosis, date of diagnosis, date of clinic appointment, physician), and deemed eligible by the RA by meeting the following criteria:

  * Age >18
  * capacity to give consent
  * has a scheduled outpatient visit (initial consult) with a palliative care provider
  * ability to speak and understand English

Exclusion Criteria:

* Not meeting the inclusion requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2018-02-26 (Actual); Study Completion 2018-02-26 (Actual)

PRIMARY OUTCOMES:
System usability as measured by the system usability scale | 1 hour
  To determine usability, the System Usability Scale will be administered to each participate. As described by usability.gov: "The participant's scores for each question are converted to a new number, added together and then multiplied by 2.5 to convert the original scores of 0-40 to 0-100. Though the scores are 0-100, these are not percentages and should be considered only in terms of their percentile ranking. Based on research, a SUS score above a 68 would be considered above average and anything below 68 is below average, however the best way to interpret the participant's results involves "normalizing" the scores to produce a percentile ranking." The original scale is a 10-item, 5-point Likert scale.

SECONDARY OUTCOMES:
Change in Palliative Care knowledge | Baseline, up to 1 hour
  Regarding the change in knowledge outcome, Two-side P value of <0.05 will infer significance. The Palliative Care Knowledge instrument is a 4-item, multiple choice assessment of palliative care knowledge. Only one answer is correct. A change in knowledge of Palliative Care will be determined based on the answer provided in the follow-up assessment
Change in Perceived Efficacy for the Patient-Physician Interaction (PEPPI) | Baseline, up to 1 hour
  Change in PEPPI will be determined using 5-point Likert response - 1 being Not at all Confident and 5 being Very Confident
Change in single-item Prepared item | Baseline, up to 1 hour
  "I feel prepared for my palliative care appointment" (5-point Likert response - Strongly Disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Kamal, MD, Principal Investigator — Duke University Health Systems
Locations (1):
- Duke University Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No